CLINICAL TRIAL: NCT03657667
Title: Evaluation of Pain Before and After Removal of Non-obstructive Kidney Stones
Acronym: ENORC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Brigham and Women's Hospital (Other); Henry Ford Health System (Other); Milton S. Hershey Medical Center (Other); Baylor Scott and White Health (Other); Indiana University (Other); University of Minnesota (Other); University of California, Davis (Other); Vanderbilt University Medical Center (Other); University of California, San Diego (Other); University of California, Los Angeles (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17.314
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Kidney Stone
Keywords: Renal Stone; Nephrolithiasis; Painful stone in kidney; Kidney stone pain
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ureteroscopy (URS) (standard treatment) (Other): Endoscopic procedure used to remove kidney stones
  Interventions: Procedure: Ureteroscopy

INTERVENTIONS:
Procedure: Ureteroscopy — Endoscopic removal of kidney stones

SUMMARY:
Pain associated with renal stone disease is typically caused by an obstructing stone that obstructs the flow of urine, which results in renal collecting system dilatation. Non-obstructing renal calculi that do not cause renal collecting system dilatation are thought to be painless. The objective of this study is to prospectively determine if the removal of non-obstructing renal calculi can reduce or eliminate participant's pain and/or improve their quality of life.

DETAILED DESCRIPTION:
Research Protocol

* Title of research project: Evaluation of pain before and after removal of non-obstructing renal calculi.
* Identification of Principal Investigator: Dr. Naeem Bhojani
* Multicentric study

Rationale & background information Renal stone disease is a common condition representing a lifetime occurrence risk of 10% in men and 7% in women. Renal stone disease is a chronic condition with a high recurrence rate. Additionally, renal stone disease is associated with considerable morbidity including pain. Pain associated with renal stone disease is typically caused by an obstructing stone that obstructs the flow of urine, which results in renal collecting system dilatation. This increases the intraluminal pressure of the urinary collecting system and stretches nerve ending in the ureteral mucosa and renal capsule. Non-obstructing renal calculi that do not cause renal collecting system dilatation are thought to be painless. There is however, some evidence that non-obstructing renal calculi located within the renal calyces actually do cause pain. In a small (n=13) retrospective study, it was found that ureteroscopic removal of non-obstructing renal calyceal stones achieved complete or partial resolution of pain in all patients. The reason for this pain is unknown.

Objective and hypothesis Objective To prospectively determine if the removal of non-obstructing renal calculi can reduce or eliminate participant's pain and/or improve their quality of life.

Hypothesis We hypothesize that the removal of non-obstructing renal calculi will decrease or eliminate the participant's pain and will improve their quality of life.

Design and methodology

Study type:

o Prospective multicentric study

Study population:

o Patients with non-obstructing renal calculi

Inclusion criteria:

* Patients with renal colic and non-obstructing renal calculi. No stone greater than 10 mm in longest diameter
* All other causes of pain have been eliminated (by clinical judgment; if the cause of pain is in doubt: assessment by a family doctor or medical specialist will be obtained)
* Patients older than 18 years old
* Moderate to severe pain (> or = 5 on BPI pain scale: pain at its worst in the last 24hrs)

Exclusion criteria:

* Patient's with anatomic abnormalities (calyceal diverticulum)
* Ureteral calculi
* Nephrocalcinosis
* Renal Tubular Acidosis (RTA), medullary sponge kidney, sarcoidosis
* Hydronephrosis or hydrocalycosis
* Minimal pain (<5 on BPI pain scale: pain at its worst in the last 24 hrs)

Methodology Our experimental plan begins with the identification of patients with non-obstructing kidney stones (< =10 mm (maximum length; measured via CT) with associated flank pain. Once all other causes of the pain have been eliminated, these patients will undergo ureteroscopy (URS) (standard treatment) to remove the offending kidney stones.

URS will be performed in the standard fashion including the use of a guide wire +/- a ureteral access sheath. Laser lithotripsy will be performed if necessary and all fragments will be extracted with the use of a basket and will be sent for stone analysis. Once the offending stone(s) has/have been removed a double J ureteral stent will be placed if deemed necessary by the surgeon. The duration of the double J ureteral stent will be determined by the surgeon.

All consented patients will undergo 3 evaluations preoperatively; The Brief Pain Inventory (BPI) (short version)[3], the Patient-Reported Outcomes Measurement Information System (PROMIS)-Pain inference/form 6b and the Wisconsin stone quality of life questionnaire (WSQOL). After removal of the renal calculi, these 3 forms will be completed by the participant at the time of stent removal or if no stent was placed, at 2 weeks post-operatively. Thereafter, the forms will be completed again at 6-8 weeks (+/- 1 week) after the initial procedure or 4 weeks (+/- 1 week) after the removal of their double J stent. Finally, the evaluations will be repeated at 12 weeks. Additionally, as with standard care at 6-8 weeks each patient will undergo post-operative imaging to determine if any renal calculi remain.

Analysis of Data With regards to the BPI, if removal of the offending kidney stone(s) is the cause of the patient's pain we expect a decrease in pain ("pain at its worst in the last 24 hours") of at least 20%. Patients included in this study should experience moderate to elevated flank pain in order to be able to detect a decrease of 20% of this pain post-intervention. This decrease will be considered clinically significant. In order to test our hypothesis, we plan to recruit a minimum of 53 patients to achieve a power of 80%. Patients will be their own control.

Sample size calculation Sample size calculation was performed using GPower software, version 3.1. Considering a baseline means Visual Analog Scale (VAS) of 7, we conservatively supposed a correlation of 0 and a standard deviation of 2.5. The standard deviation was estimated with the range (i.e. σ ≈ range/4), assuming the VAS to be normally distributed. Thus, a sample size of n = 53 is required to ensure at least 80% power to detect a clinically significant difference of 20 % (post-mean = 5.6), at a significance level of 5 %.

Impact of the Proposed Research The results of this study will conceivably provide significant evidence on whether small non-obstructing renal calculi can cause flank pain.

Ethical considerations

* All personal identifiers, such as patients' names, will be removed and replaced with a unique numerical code.
* Only the principal investigator and approved study staff will be able to identify the patients and have access to the study files.
* The consent will be kept in a locked office at the Research Center of the University of Montéral Hospital Center (CRCHUM).
* The data collected will be protected in files with a password on secure servers (computers).
* The data will be kept during a period of 10 years on secured computers with passwords by the principal investigator of this research project at the CRCHUM. After that, they will be destroyed.
* The combined results from this study may be used to prepare reports and summaries for scientific publications and presentations at scientific meetings. If they are, identity of the patients will remain confidential.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal colic and non-obstructing renal calculi. No stone greater than 10 mm in longest diameter
* All other causes of pain have been eliminated (by clinical judgment; if the cause of pain is in doubt: assessment by a family doctor or medical specialist will be obtained)
* Patients older than 18 years old
* Moderate to severe pain (> or = 5 on BPI pain scale: pain at its worst in the last 24hrs)

Exclusion Criteria:

* Patient's with anatomic abnormalities (calyceal diverticulum)
* Ureteral calculi
* Nephrocalcinosis
* RTA, medullary sponge kidney, sarcoidosis
* Hydronephrosis or hydrocalycosis
* Minimal pain (<5 on BPI pain scale: pain at its worst in the last 24 hrs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | 12 weeks
  evaluated using The Brief Pain Inventory; scale from 0-10; worst pain is 10

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Bhojani, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (9):
- United States (8):
  - University of California, Davis, Davis, California
  - University of California, San Diego, San Diego, California
  - Indiana University, Bloomington, Indiana
  - Brigham And Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Health, Temple, Texas
- Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Travaglini F, Bartoletti R, Gacci M, Rizzo M. Pathophysiology of reno-ureteral colic. Urol Int. 2004;72 Suppl 1:20-3. doi: 10.1159/000076586. PMID 15133328
- [Result] Jura YH, Lahey S, Eisner BH, Dretler SP. Ureteroscopic treatment of patients with small, painful, non-obstructing renal stones: the small stone syndrome. Clin Nephrol. 2013 Jan;79(1):45-9. doi: 10.5414/CN107637. PMID 23006342
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Penniston KL, Antonelli JA, Viprakasit DP, Averch TD, Sivalingam S, Sur RL, Pais VM Jr, Chew BH, Bird VG, Nakada SY. Validation and Reliability of the Wisconsin Stone Quality of Life Questionnaire. J Urol. 2017 May;197(5):1280-1288. doi: 10.1016/j.juro.2016.11.097. Epub 2016 Nov 23. PMID 27889419
- [Result] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Result] Farrar JT, Portenoy RK, Berlin JA, Kinman JL, Strom BL. Defining the clinically important difference in pain outcome measures. Pain. 2000 Dec 1;88(3):287-294. doi: 10.1016/S0304-3959(00)00339-0. PMID 11068116
- [Result] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Result] Hozo SP, Djulbegovic B, Hozo I. Estimating the mean and variance from the median, range, and the size of a sample. BMC Med Res Methodol. 2005 Apr 20;5:13. doi: 10.1186/1471-2288-5-13. PMID 15840177